CLINICAL TRIAL: NCT01562340
Title: A Pilot Trial Assessing the Effect of Pomegranate Juice and Extract on Biomarkers of Oxidative Stress, Systemic Inflammation, and Monocyte Function in Hemodialysis Patients
Brief Title: Pomegranate and Hemodialysis Pilot Trial
Acronym: POM Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 41986-D
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: End Stage Renal Disease; Cardiovascular Disease; Inflammation
Keywords: Hemodialysis; End stage renal disease; Oxidative stress; Inflammation; Endothelial dysfunction; Cardiovascular disease; Antioxidants; Flavonoids
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases; Inflammation | interventions — pomegranate fruit rind

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate fruit extract (Active Comparator)
  Interventions: Other: Pomegranate fruit extract
- Pomegranate juice (Active Comparator)
  Interventions: Other: Pomegranate juice

INTERVENTIONS:
Other: Pomegranate juice — Pomegranate juice (100 mL) 3 times per week (taken prior to hemodialysis session) for 4 weeks. Followed by 4 week wash-out (no intervention), then crossover to Comparator arm.
  Other Names: Research Juice 100%
  Arms: Pomegranate juice
Other: Pomegranate fruit extract — Pomegranate fruit extract in single capsule (1050 mg) daily by mouth for 4 weeks. Followed by 4 week wash-out (no intervention), then crossover to Comparator arm.
  Other Names: Clinical Active POMxp
  Arms: Pomegranate fruit extract

SUMMARY:
In this study, the investigators will administer pomegranate juice or fruit extract as a targeted antioxidant therapy to hemodialysis patients.

The investigators will examine whether these pomegranate products will be safe and well-tolerated. The investigators will also examine whether these products may lead to improvements in blood serum biomarkers of:

* oxidative stress status
* inflammatory status
* endothelial dysfunction

DETAILED DESCRIPTION:
There are currently more than 400,000 patients receiving chronic dialysis therapy in the United States. Cardiovascular and infectious diseases are the leading causes of death in hemodialysis patients, accounting for over 50% of all-cause mortality.

There is a complex interaction of inflammation, oxidative stress, and endothelial dysfunction in contributing to cardiovascular and infectious risk in dialysis patients. Since there is much evidence that an increase in oxidative stress contributes to risk of disease in dialysis patients, it is logical to hypothesize the antioxidant therapy may be beneficial in reducing these risks.

In addition to vitamins C and E, the most common and active antioxidant compounds that occur naturally in foods are flavonoids. Dietary flavonoids are highly bioavailable, and have been shown to confer antioxidant protection, inhibit platelet activation, exert vasorelaxant effects, and reduce inflammation in human studies. In animal model studies, dietary flavonoids have been shown to reduce the development of atherosclerosis. Polyphenols also have potent antibacterial, antifungal, and antiviral activities.

Pomegranate juice is a rich source of potent phenolic antioxidants, which have been demonstrated to have anti-atherogenic and vasorelaxant properties. Pomegranate derived polyphenols have also been demonstrated to inhibit platelet activation.

Although available data are limited, several studies suggest that dietary phenols may have beneficial effects in patients undergoing dialysis treatment. These include improvements in lipoprotein profiles, reductions in circulating inflammatory and oxidative stress biomarkers, reductions in infectious complications, and improvements in inflammatory biomarkers. These observations, though limited, suggest that polyphenol based supplementation strategies may be effective in reducing complications in those undergoing dialysis treatment.

In this study, the investigators will administer pomegranate juice and/or fruit extract as a targeted antioxidant therapy. The investigators will examine whether these pomegranate products will be safe and well-tolerated. The investigators will also examine whether these products may lead to improvements in biomarkers of oxidative stress status, inflammatory status, and endothelial dysfunction in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease receiving thrice weekly hemodialysis
* Age > 18 or < 85 years
* Life expectancy greater than one year
* Ability to understand and provide informed consent for participation in the study

Exclusion Criteria:

* History of poor adherence to hemodialysis or medical regimen
* Prisoners, patients with significant mental illness, and other vulnerable populations
* AIDS (HIV seropositivity is not an exclusion criteria)
* Active malignancy excluding basal cell carcinoma of the skin
* Gastrointestinal dysfunction requiring parenteral nutrition
* History of functional kidney transplant < 6 months prior to study entry
* Anticipated live donor kidney transplant
* Patients taking vitamin E supplements > 60 IU/day, vitamin C > 150 mg/day or other antioxidant or nutritional supplements
* Incident hemodialysis patients (defined as within 30 days of dialysis initiation)
* Patients hospitalized for more than 5 days within the past 30 days.
* Patients with a history of a major atherosclerotic event (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery, and stroke) within three months
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Markers of oxidative stress | 12 weeks
  Oxidative stress: F2-isoprostanes
Markers of inflammation | 12 weeks
  Inflammation: C-reactive protein, Interleukin-6, and white blood cell count
Markers of endothelial function | 12 weeks
  Endothelial function: Monocyte functional assays (cytokines)

SECONDARY OUTCOMES:
Number of subjects with adverse events and type of event | 12 weeks
  Adverse reactions to pomegranate juice
  Adverse reactions to pomegranate fruit extract

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (1):
- Northwest Kidney Centers, Seattle, Washington, United States

REFERENCES:
- [Derived] Rivara MB, Mehrotra R, Linke L, Ruzinski J, Ikizler TA, Himmelfarb J. A pilot randomized crossover trial assessing the safety and short-term effects of pomegranate supplementation in hemodialysis patients. J Ren Nutr. 2015 Jan;25(1):40-9. doi: 10.1053/j.jrn.2014.07.006. Epub 2014 Sep 11. PMID 25218876
- See also: Kidney Research Institute at the University of Washington — http://kri.washington.edu/
- See also: Northwest Kidney Centers — http://nwkidney.org